CLINICAL TRIAL: NCT01402752
Title: System for Measuring Non-invasive Blood Flow in the Tracheobronchial Mucosa: Validation of Reproducibility
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: 20131209 Regulatory authorization is currently blocked at the ANSM.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2011/CLM-02
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): All patients included in this study according to stated inclusion and exclusion criteria.
  Interventions: Biological: Blood flow to the tracheo-bronchial mucosa

INTERVENTIONS:
Biological: Blood flow to the tracheo-bronchial mucosa — Measurement of blood flow to the tracheo-bronchial mucosa via differential absorption of diluted dimethyl ether tracer gas.

SUMMARY:
The primary objective of this study is to evaluate the reproducibility of a method of measuring blood flow rates to the tracheo-bronchial mucosa using diluted dimethyl ether as a tracer.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan

Exclusion Criteria:

* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Patient is pregnant
* Patient is breast feeding
* The patient is a smoker
* The patient has, or has a history of, chronic respiratory insufficiency
* The patient has a contra-indication for a treatment necessary in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The reproducibility of two measures of Qaw at a five minute interval | Five minutes
  Qaw is the blood flow measured in the tracheobronchial mucosa. Qaw = VDME/(FDME*alpha*10s) where VDME is the volume of dimethyl-ether exhaled (ml), FDME is the mean concentration of dimethyl-ether (%), alpha is the Bunsen coefficient for the dissolution of dimethyl ether in tissues and blood at 37°C (i.e. 9ml/ml).

SECONDARY OUTCOMES:
The time necessary to complete one measure of Qaw (minutes) | Day 1
  Qaw = blood flow measured in the tracheobronchial mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Charles Le Merre, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes